CLINICAL TRIAL: NCT03113123
Title: Prevention of HIV in "Île-de-France"
Acronym: ANRS-PREVENIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS PREVENIR; 2016-A01577-44 (Registry Identifier: French Drug Regulatory Authorities Clinical Trial System)
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: HIV Infections
Keywords: Adherence; Prevention; Tenofovir; Emtricitabine; Antiretroviral; Prophylaxis; Men who have sex with men
MeSH Terms: conditions — HIV Infections; Homosexuality | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEP with Truvada® (Other): On demand PrEP (only for MSM - with the possibility of dosing schedule switching): 2 pills of Truvada within 24 to 2 hours prior first sexual intercourse, then 1 pill every 24 hours during the period of sexual activity with one pill after the last sexual intercourse, and one last pill 24 hours later
  Continuous PrEP: 1 pill every 24 hours, at least 7 days before the first sexual intercourse. When PrEP is to be discontinued, 2 pills 24 hours apart after the last sexual intercourse then stop PrEP. If PrEP is to be resumed, 1 pill every 24 hours, started at least 7 days before the first sexual intercourse or 2 pills at least 2 hours before the first sexual intercourse and then 1 pill every 24 hours.
  Interventions: Drug: PrEP with Truvada®

INTERVENTIONS:
Drug: PrEP with Truvada® — Associated with:
  * STD screening/treatment for syphilis, gonorrhoea and chlamydiae
  * HIV screening/therapy
  * Questionnaire
  * Addiction, social or psychological follow-up care if needed
  * Peer interactive counselling (peer counselors/nurses/physicians experienced with therapeutic education) at the baseline visit and at every follow-up visit up to 6 months. After 6 months, counselling will be provided at the request of participants if they need it. Counselors will remain in contact with the participants between visit to answer any questions relative to PrEP, treatment and prevention, and to facilitate participants interactions with study sites.
  Other Names: Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC)

SUMMARY:
Interventional HIV prevention strategy based on pre-exposure prophylaxis (PrEP) with Truvada® for people in the Île-de-France area (or Paris region) who don't have HIV but who are at high risk of becoming infected with HIV (men who have sex with men (MSM), transgender men and women, heterosexual men and women, sex workers, migrants) in combination with overall prevention services (communautary-based or educational counselling; addiction, social and psychological care; condoms and lubricating gel; clean injection equipment; sexually transmitted diseases (STD) screening and treatment; hepatitis A virus (HAV), hepatitis B virus (HBV) and hepatitis C virus (HCV) vaccinations and post-exposure treatment of HIV infection as soon as possible after diagnosis using an antiretroviral combination recommended by the French Guidelines on HIV treatment).

The individual benefit being already demonstrated in clinical trials, the aim is to demonstrate the public health impact of the interventional HIV prevention strategy by reducing the risk of getting HIV-1 infection of at least 15% of new diagnosis of HIV infections among MSM/transgender in the Ile-de-France area after a 3-year period.

DETAILED DESCRIPTION:
Assuming the PrEP efficacy of 80% and that 85% of included participants being MSM - the objective is to evidence a decrease of at least 15% of new diagnosis of HIV infections among MSM in Ile-de-France area. This objective is in the framework of a commitment of large cities against AIDS with the political support of the City of Paris for the "Paris sans SIDA" program and the commitment of the Île-de-France area.

Secondary Objectives:

* Prevalence of HIV infection at the screening visit (undiagnosed epidemic)
* Incidence of HIV infection according to back-calculation approach, and by key subgroups

Operational Objectives:

* Evaluate the origin of the recruitment according to the risk groups and the outreach actions
* Assess linkage to care for PrEP, retention in the study, reasons for consent withdrawal and satisfaction of the participants according to the screening site, the type of PrEP supply, the costs of global care, the key subgroups, the type of counselling, the time from STD testing to initiation of PrEP treatment in study sites
* Impact of a less intense counselling than the one provided in the ANRS IPERGAY trial, on adherence and efficacy of PrEP by comparing the incidence observed in MSM enrolled in the current study to that evidenced in the ANRS IPERGAY trial, with a method similar to that used in the Partner demonstration project in Kenya and Uganda.
* Impact of the communautary-based and educational counselling

Clinical Objectives:

* Estimation, in individuals seeking for PrEP and thus getting tested for HIV infection, the prevalence of HIV infection in different key subgroups, which is a surrogate marker of the undiagnosed (or "hidden") epidemic
* Evaluate who will become HIV-infected during the course of the study while on PrEP, the proportion of patients on combined antiretroviral treatment and the proposition of patients with a suppressed HIV viral load 12 months after HIV infection
* Evaluate the participants' need for post-exposure prophylaxis during the course of the study
* Adherence to PrEP (questionnaire and dried blood spots)
* Assessment of the PrEP dosing schedule used by MSM participants (daily or intermittent) throughout the course of the study
* Assessment of PrEP tolerability and safety
* Comprehensive study of incident HIV infections in those on PrEP (incidence, emergence of drug-associated resistance mutations, adherence to PrEP at the closest visit before HIV seroconversion and at previous visits)

Participants Behavior:

* Acceptability of PrEP (including those who will decline participation in the study) and during the course of the study, and retention in the study.
* Impact of PrEP, within a comprehensive prevention offer, on sexual behavior of the participants throughout follow-up
* Factors associated with the integration of PrEP in the daily routine of participants:

  * Qualitative study to explore the motivations, difficulties, behavior and expectations of the participants, their knowledge and communication on their use of PrEP
  * Reasons related to the choice of the prevention strategy used in terms of dosing schedule (continuous or on demand in MSM) and type of counselling and participation to focus groups.

Care Providers Behavior: Evaluation of knowledge, beliefs, perception and practice of the physicians, nurse and peer counselors involved in delivery of PrEP in the study

Social epidemiology: Evaluation of social and/or territorial inequalities and disparities

Cost-effectiveness of the comprehensive prevention strategy

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Men/transgender men/women who have sex with men, heterosexual men and women, sex workers
* Negative for HIV-1 and HIV-2 (with a fourth generation enzyme-linked immunosorbent assay (ELISA) assay)
* Willing the geocoding of the postal address and to be contacted via telephone or email, on a regular basis
* Willing to comply to visits schedule (every 3 months)
* Health security program
* Informed consent form signed
* High risk of acquiring HIV infection:

  * For MSM and transgenders:

    * Anal sex with at least two different sexual partners and no consistent condom use over the last 6 months
    * And/or history of STD during the last 12 months (syphilis, gonorrhea , chlamydiae, HBV or HCV infection)
    * And/or history of non-occupational post-exposure prophylaxis (PEP) during the last 12 months
    * And/or using psycho-actives drugs during sexual intercourses (cocaine, gammahydroxybutyric acid (GHB), Methylenedioxymethamphetamine (MDMA), mephedrone)
    * And/or having an HIV-infected sexual partner with a detectable plasma viral load (> 50 copies (cp)/milliliter (ml))
  * For heterosexual:

    * Sexual intercourse with 1 partner originating from regions with high prevalence of HIV infection (> 1%) (South America, Sub-Saharan Africa, South-East Asia, Eastern Europe, French Guyana) and no consistent condom use
    * and/or sex workers
    * and/or having a sexual partner who is an intravenous drug users sharing injection material
    * and/or having an HIV-infected sexual partner with a detectable plasma viral load (> 50 cp/ml)

Exclusion Criteria:

* Stable and exclusive relationship with an HIV-negative partner, or with an HIV-positive partner on antiretroviral therapy (ART) with a plasma viral load < 50 cp/ml
* Positive HIV infection
* Clinical signs of positive HIV infection
* Consistent condom use during sexual intercourse
* Expected trip abroad for 3 consecutive months
* Creatinine clearance lower than 50ml/min
* History of chronic renal disease, osteoporosis or osteopenia
* Receiving an investigational drug
* Receiving or will receive potentially nephrotoxic treatments
* Gastro-intestinal condition that could limit drug absorption
* Potentially non compliant participants
* Breastfeeding
* Hypersensitivity to TDF/FTC
* Positive HBs antigen or isolated anti hepatitis B core (HBc) antibodies if not willing to take daily PrEP
* Severe condition (lymphoma, other cancers, cardio-vascular disease, end-stage renal failure, uncontrolled diabetes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3257 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2024-05-02 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of new HIV diagnosis | three years
  Number of new HIV infections

SECONDARY OUTCOMES:
Number of recent infections | three years
  Impact of the study on the total number and on recent HIV infections in Île-de- France, and in each key subgroup
Prevalence of HIV-infection at the screening visit (undiagnosed epidemic) | two years
  Number of HIV-infected persons at screening visit
Incidence of HIV infection | three years
  Incidence of HIV infection in Paris and in the Île-de-France area according to back-calculation approach, and by key subgroups (MSM, transgenders, migrants, etc.)
Retention in the study | two years
  Retention in the study, reasons for consent withdrawal
Counselling | three years
  Impact of a less intense counselling than the one provided in the ANRS IPERGAY trial, on adherence and efficacy of PrEP
Type of counselling | three years
  Impact of counselling according to the type of counselling provided: communautary-based or educational
Post-exposure prophylaxis | three years
  Evaluate the participants' need for post-exposure prophylaxis during the course of the study
Adherence to PrEP | three years
  Evaluation of adherence by self-administered online questionnaires on last sexual intercourse
  * Questionnaire on the use of PrEP during the last month prioir to study visit
  * Dried blood spots to assess TVF-DP and/or FTC-TP in red cells
PrEP dosing schedule | three years
  Assessment of the PrEP dosing schedule used by MSM participants (daily or intermittent) throughout the course of the study
Safety and tolerability | three years
  Assessment of PrEP tolerability and safety particularly: incidence of drug-related adverse events, incidence of grade 3-4 adverse events, incidence of adverse events leading to PrEP discontinuation
Incident HIV infections | three years
  Comprehensive study of incident HIV infections in those on PrEP Incidence of HIV-infection on PrEP
  * Emergence of drug-associated resistance mutations (in particular FTC and tenofovir- mutations at positions 184, 65, and 70 in reverse transcriptase gene)
  * Adherence to PrEP at the closest visit before HIV seroconversion and at previous visits
Participants Behavior | three years
  Acceptability of PrEP (including those who will decline participation in the study) and during the course of the study.
  Impact of PrEP, within a comprehensive prevention offer, on sexual behavior of the participants throughout follow-up
  * Number of partners during the previous 2 months
  * Number of sexual intercourses during the previous 4 weeks
  * Use of condom at last sexual intercourse
  * Incidence of STIs
Integration of PrEP in the daily routine of participants | three years
  * Factors associated with the integration of PrEP in the daily routine of participants
    - Qualitative study to explore the motivations, difficulties, behavior and expectations of the participants, their knowledge and communication on their use of PrEP. We will focus on:
  * Change in the use of sexual networks (internet, sex clubs, backrooms, sauna)
  * Feeling of sexual well-being during sexual intercourse (less worried about getting HIV infection)
  * Condom use (withdrawal of condom use)
Care Providers Behavior | three years
  Evaluation of knowledge, beliefs, perception and practice of the physicians, nurse and peer counselors involved in delivery of PrEP in the study
Social epidemiology | three years
  * Evaluation of social and/or territorial inequalities and disparities through collection of relevant indicators
  * Socio-economic status
  * Social insertion: marital status etc.
  * Origin (according to Ined definition) : french, french born from immigrant parents, immigrants
  * Précar score
  * Socio-economical background (according to IRIS indicator)
Cost-effectiveness | three years
  Cost-effectiveness of the comprehensive prevention strategy provided in this study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel MOLINA, Pr, Principal Investigator — Hôpital Saint Louis, Paris, FRANCE; Jade GHOSN, MD, Study Chair — Hôpital Hôtel-Dieu, Paris, FRANCE
Locations (21):
- France (21):
  - Hôpital Avicenne, Bobigny
  - Hôpital Jean Verdier, Bondy
  - Hôpital Ambroise-Paré, Boulogne
  - Hôpital Antoine Béclère, Clamart
  - Hôpital Louis Mourier, Colombes
  - Hôpital Henry Mondor, Créteil
  - Hôpital Raymond Poincaré, Garches
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Marc Jacquet, Melun
  - Hôpital Cochin, Paris
  - Hôpital Hôtel Dieu, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Bichat-Claude-Bernard, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - CHI Poissy Saint Germain en Laye, Saint-Germain-en-Laye
  - Hôpital Foch, Suresnes
  - Hôpital André Mignot, Versailles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Protiere C, Sagaon-Teyssier L, Donadille C, Sow A, Gaubert G, Girard G, Mora M, Assoumou L, Beniguel L, Michels D, Ghosn J, Costagliola D, Rojas Castro D, Molina JM, Spire B; ANRS PREVENIR Study-Group. Perception of PrEP-related stigma in PrEP users: Results from the ANRS-PREVENIR cohort. HIV Med. 2023 Aug;24(8):938-945. doi: 10.1111/hiv.13491. Epub 2023 Apr 12. PMID 37046178
- [Derived] Molina JM, Ghosn J, Assoumou L, Delaugerre C, Algarte-Genin M, Pialoux G, Katlama C, Slama L, Liegeon G, Beniguel L, Ohayon M, Mouhim H, Goldwirt L, Spire B, Loze B, Surgers L, Pavie J, Lourenco J, Ben-Mechlia M, Le Mestre S, Rojas-Castro D, Costagliola D; ANRS PREVENIR Study Group. Daily and on-demand HIV pre-exposure prophylaxis with emtricitabine and tenofovir disoproxil (ANRS PREVENIR): a prospective observational cohort study. Lancet HIV. 2022 Aug;9(8):e554-e562. doi: 10.1016/S2352-3018(22)00133-3. Epub 2022 Jun 27. PMID 35772417
- See also: sponsor of the study — http://www.anrs.fr